CLINICAL TRIAL: NCT01462292
Title: An Exploratory Study to Assess Two Doses of GSK2402968 in the Treatment of Ambulant Boys With Duchenne Muscular Dystrophy
Brief Title: A Clinical Study to Assess Two Doses of GSK2402968 in Subjects With Duchenne Muscular Dystrophy (DMD)
Acronym: DMD114876
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114876
Record Dates: First submitted 2011-10-03; First posted 2011-10-31 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-08

CONDITIONS: Muscular Dystrophies
Keywords: 968; Duchenne Muscular Dystrophy; GSK2402968; DMD; Duchenne; GSK
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GSK2402968 3 mg/kg/week (Experimental): 3 mg/kg/week of investigational product
  Interventions: Drug: GSK2402968 3mg/kg/week
- GSK2402968 6 mg/kg/week (Experimental): 6 mg/kg/week of investigational Product
  Interventions: Drug: GSK2402968 6 mg/kg/week
- Placebo to match GSK2402968 3 mg/kg/week (Experimental): Placebo
  Interventions: Drug: Placebo to match GSK2402968 3 mg/kg/week
- Placebo to match GSK2402968 6 mg/kg/week (Experimental): Placebo
  Interventions: Drug: Placebo to match GSK2402968 6 mg/kg/week

INTERVENTIONS:
Drug: GSK2402968 3mg/kg/week — Comparison of 2 doses of GSK2402968
  Arms: GSK2402968 3 mg/kg/week
Drug: GSK2402968 6 mg/kg/week — Comparison of 2 doses of GSK2402968
  Arms: GSK2402968 6 mg/kg/week
Drug: Placebo to match GSK2402968 3 mg/kg/week — Matched placebo
  Arms: Placebo to match GSK2402968 3 mg/kg/week
Drug: Placebo to match GSK2402968 6 mg/kg/week — Matched Placebo
  Arms: Placebo to match GSK2402968 6 mg/kg/week

SUMMARY:
The purpose of this study is to determine if GSK2402968 is effective in the treatment of ambulant boys with Duchenne muscular dystrophy resulting from a mutation thought to be corrected by exon 51 skipping. Two doses of GSK2402968 and placebo will be used in this study.

DETAILED DESCRIPTION:
Boys with Duchenne Muscular Dystrophy (DMD) suffer from a relentless, progressive and fatal disease due to lack of dystrophin, a critical muscle protein. There is currently no known cure for the disease. GSK2402968 is thought to correct several genetic mutations through skipping of exon 51 and therefore targets only those boys with these mutations.

A reasonable hypothesis is that increasing dystrophin will result in clinical improvement, and that the amount of dystrophin expressed will correlate with clinical improvement above a threshold level (e.g. around 30% of control). The initial limited efficacy data from completed and ongoing unblinded studies with GSK2402968 are encouraging as they have demonstrated de novo production of dystrophin and improved walking ability (primary efficacy endpoint) after 48 weeks of treatment which has been generally well tolerated.

This study is designed to explore the efficacy, safety and pharmacokinetics of two doses of GSK2402968 given over 24 weeks. The two doses to be assessed are 6mg/kg/week and 3mg/kg/week. Based on pharmacokinetic and pharmacodynamic modeling, it is predicted at steady-state that the 6 mg/kg/week dose will induce dystrophin expression greater than 30% of control. The 3 mg/kg/week dose was chosen as modeling predicts 3 mg/kg/week of GSK2402968 will produce dystrophin expression in the range of 18-22%. Potential variability between subjects could theoretically produce higher expression and lead to a dystrophin level correlated with clinical improvement.

Following the treatment period, the study has a 24 week post-treatment phase. The purpose of the post-treatment phase is to model the half-life of dystrophin, assess maintenance of response, and provide information about resolution of adverse event and laboratory abnormalities following cessation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ambulant subjects with Duchenne muscular dystrophy (DMD) resulting from a mutation/deletion within the DMD gene, confirmed by a state-of-the-art DNA diagnostic technique covering all DMD gene exons, including but not limited to MLPA (Multiplex Ligation-dependent Probe Amplification), CGH (Comparative Genomic Hybridisation), SCAIP (Single Condition Amplification/Internal Primer) or H-RMCA (High-Resolution Melting Curve Analysis), and correctable by GSK2402968-induced DMD exon 51 skipping
* Males, aged at least 5 years,
* Life expectancy of at least 1 year,
* Able to rise from floor in < or =15 seconds (without aids/orthoses) at Screening Visit 1 and Screening Visit 2,
* Able to complete 6 Minute Walk Distance (6MWD) test with minimal distance of at least 75 meters, with reproducible results (within 20% of each other) at Screening Visit 1, Screening Visit 2 and at the baseline visit prior to randomization,
* Receiving oral glucocorticoids for a minimum of 6 months immediately prior to screening, with no significant change in total daily dosage or dosing regimen for a minimum of 3 months immediately prior to screening and a reasonable expectation that total daily dosage and dosing regimen will not change significantly for the 48 week duration of the study (Dose adjustments that are based on weight changes are permitted),
* QTc <450msec (based on single or average QTc value of triplicate ECGs obtained over a brief recording period), or <480 msec for subjects with Bundle Branch Block. Note: QTc may be either QTcB or QTcF, and machine read or manual overread
* Willing and able to comply with all protocol requirements and procedures,
* Able to give informed assent and/or consent in writing signed by the subject and/or parent(s)/legal guardian (according to local regulations).

Exclusion Criteria:

* Any additional missing exon for DMD that cannot be treated with GSK2402968,
* Current or history of liver disease or impairment including :

  1. an INR vaue above 1.5 is in and of itself exclusionary
  2. a total bilirubin greater than 2 times the Upper Limit of Normal is in and of itself exclusionary
  3. a GGT greater than 2 times the Upper Limit of Normal is in and of itself exclusionary
* Current or history of renal disease or impairment,
* Baseline platelet count below the Lower Limit of Normal,
* aPPT above the Upper Limit of Normal,
* History of significant medical disorder which may confound the interpretation of either efficacy or safety data e.g. inflammatory disease
* Acute illness within 4 weeks of the first anticipated administration of study medication which may interfere with study assessments,
* Use of anticoagulants, antithrombotics or antiplatelet agents, previous treatment with investigational drugs, idebenone or other forms of Coenzyme Q10 within 1 month of the first administration of study medication,
* Current or anticipated participation in any investigational clinical studies,
* Positive hepatitis B surface antigen, hepatitis C antibody test (if verified via RIBA or PCA testing), or human immunodeficiency virus (HIV) test at screening,
* Symptomatic cardiomyopathy. If subject has a left ventricular ejection fraction <45% at Screening, the investigator should discuss inclusion of subject in the study with the medical monitor,
* Children in Care. The definition of a Child in Care is a child who has been placed under the control or protection of an agency, organisation, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation. The definition of a child in care can include a child cared for by foster parents or living in a care home or institution, provided that the arrangement falls within the definition above. The definition of a child in care does not include a child who is adopted or has an appointed legal guardian

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-10-26 (Actual); Primary Completion 2013-05-21 (Actual); Study Completion 2013-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- United States (14):
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Gulf Breeze, Florida
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 51 male participants, with Duchenne Muscular Dystrophy were randomized in the study. The study was conducted from 26 October 2011 to 04 November 2013.
Groups:
- Placebo (Combined): The participants in this arm were administered matching placebo subcutaneously for 24 Weeks. It was provided as 3 milliliter (mL) vials containing 1 mL sterile solution.
- GSK2402968 3 mg/kg/Week: The participants in this arm were administered with 3 milligram (mg) per kilogram (kg) GSK2402968, subcutaneously for 24 weeks. It was provided as 3 mL vials containing 1 mL sterile solution. The concentration of drisapersen solution was 200 mg/mL
- GSK2402968 6 mg/kg/Week: The participants in this arm were administered with 6 mg per kg GSK2402968, subcutaneously for 24 weeks. It was provided as 3 mL vials containing 1 mL sterile solution. The concentration of drisapersen solution was 200 mg/mL
Period: Overall Study
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Started | 16 | 17 | 18
Completed | 16 | 17 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo (Combined): The participants in this arm were administered matching placebo subcutaneously for 24 Weeks. It was provided as 3 mL vials containing 1 mL sterile solution.
- GSK2402968 3 mg/kg/Week: The participants in this arm were administered with 3 mg per kilogram kg GSK2402968, subcutaneously for 24 weeks. It was provided as 3 mL vials containing 1 mL sterile solution. The concentration of drisapersen solution was 200 mg/mL.
- Total: Total of all reporting groups
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week | Total
Number analyzed (Participants) | 16 | 17 | 18 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.0 (1.79) | 7.8 (1.91) | 7.6 (2.70) | 7.8 (2.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 16 | 17 | 18 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 14 | 16 | 15 | 45
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Muscle Function Using the 6 Minute Walking Distance
Description: The participants during this assessment were asked to walk, at their own preferred speed, up and down a fixed distance until they were told to stop after 6 minutes. The participants were warned of the time and were told to stop earlier if they feel unable to continue. The total distance walked within the duration of 6 minutes (or until the participant stopped in case of early termination of the test), was recorded in meters. Change from Baseline, was defined as the post-randomization value minus the Baseline value. Baseline was defined as Week 0.
Time Frame: Baseline (Week 0) and Week 24
Population: Intent to Treat (ITT) Population was defined as all participants who were randomized to the study, received at least one dose of study medication and have at least one post-Baseline efficacy assessment
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 16 | 17 | 18
Meters | -10.98 (10.666) | -19.93 (9.964) | 16.12 (9.941)
Statistical Analysis 1: Comparison: Placebo (Combined) vs GSK2402968 3 mg/kg/Week; Treatment difference: Placebo Vs GSK2402968 3 mg; Test type: Superiority or Other; p = 0.554, Mixed Model Repeated Measures — Due to the two comparisons for the two different doses, the type 1 error rate (5% overall) was preserved by utilizing a hierarchical approach, testing the 6mg/kg GSK2402968 dose first; Model included terms for treatment, visit, treatment by visit, centre grouping, baseline and baseline by visit; Mean Difference (Net) = -8.946, 95% CI 2-sided [-39.122 to 21.229]
Statistical Analysis 2: Comparison: Placebo (Combined) vs GSK2402968 6 mg/kg/Week; Treatment difference: Placebo Vs GSK2402968 6 mg; Test type: Superiority or Other; p = 0.069, Mixed Model Repeated Measures — Due to the two comparisons for the two different doses, the type 1 error rate (5% overall) was preserved by utilising a hierarchical approach, testing the 6mg/kg GSK2402968 dose first; Model included terms for treatment, visit, treatment by visit, centre grouping, baseline and baseline by visit; Mean Difference (Net) = 27.099, 95% CI 2-sided [-2.210 to 56.408]

2. Secondary Outcome: Change From Baseline in Rise From Floor Time at Week 24
Description: The rise from floor was assessed, when the participants stood from a standardized supine position as quickly as possible when told to go. Time was recorded with a stopwatch from the initiation of movement until the assumption of upright standing. No aids or orthoses were allowed. Change from Baseline, was defined as the post-randomization value minus the Baseline value. Baseline was defined as Week 0.
Time Frame: Baseline (Week 0) and Week 24
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 16 | 17 | 18
Seconds | 1.12 (0.700) | 1.50 (0.662) | 1.95 (0.656)
Statistical Analysis 1: Comparison: Placebo (Combined) vs GSK2402968 3 mg/kg/Week; Treatment difference: Placebo Vs GSK2402968 3 mg; Test type: Superiority or Other; p = 0.699, ANCOVA — No adjustment for multiplicity was made, so p-values should not be used to make conclusions with regards to statistical significance; Model included terms for treatment, centre grouping and baseline; Mean Difference (Net) = 0.387, 95% CI 2-sided [-1.618 to 2.392]
Statistical Analysis 2: Comparison: Placebo (Combined) vs GSK2402968 6 mg/kg/Week; Treatment difference: Placebo Vs GSK2402968 6 mg; Test type: Superiority or Other; p = 0.384, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Model included terms for treatment, centre grouping and baseline; Mean Difference (Net) = 0.831, 95% CI 2-sided [-1.072 to 2.735]

3. Secondary Outcome: Change From Baseline in 4 Stair Climb Ascent/Descent Time at Week 24
Description: During this assessment, the participants were asked to ascend and descend four steps. The time for this was recorded with a stopwatch from the initiation of movement until the participant stands on the fourth step, (going up and going down separately). A flight of steps with handrail were used for this test. Change from Baseline, was defined as the post-randomization value minus the Baseline value. Baseline was defined as Week 0.
Time Frame: Baseline (Week 0) and Week 24
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 16 | 17 | 18
seconds
  Ascent time | 0.59 (0.308) | 0.59 (0.295) | -0.22 (0.295)
  Descent time | 0.60 (0.473) | -0.09 (0.442) | 0.19 (0.440)
Statistical Analysis 1: Comparison: Placebo (Combined) vs GSK2402968 3 mg/kg/Week; Placebo (combined) Vs GSK2402968 3 mg/kg/week, Ascent Week 24; Test type: Superiority or Other; p = 0.997, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Model included terms for treatment,centre grouping and baseline; Mean Difference (Net) = 0.002, 95% CI 2-sided [-0.883 to 0.886]
Statistical Analysis 2: Comparison: Placebo (Combined) vs GSK2402968 6 mg/kg/Week; Placebo (combined) Vs GSK2402968 6 mg/kg/week, Ascent, Week 24; Test type: Superiority or Other; p = 0.064, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Model included terms for treatment, centre grouping and baseline; Mean Difference (Net) = -0.803, 95% CI 2-sided [-1.655 to 0.048]
Statistical Analysis 3: Comparison: Placebo (Combined) vs GSK2402968 3 mg/kg/Week; Placebo (combined) Vs GSK2402968 3 mg/kg/week, Descent Week 24; Test type: Superiority or Other; p = 0.311, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Model included terms for treatment, centre grouping and baseline; Mean Difference (Net) = -0.685, 95% CI 2-sided [-2.033 to 0.662]
Statistical Analysis 4: Comparison: Placebo (Combined) vs GSK2402968 6 mg/kg/Week; Placebo (combined) Vs GSK2402968 6 mg/kg/week, Descent Week 24; Test type: Superiority or Other; p = 0.523, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Model included terms for treatment, centre grouping and baseline; Mean Difference (Net) = -0.412, 95% CI 2-sided [-1.702 to 0.878]

4. Secondary Outcome: Change From Baseline in 10 Meter Walk/Run at Week 24
Description: The participants during this assessment were asked to traverse marked 10-meter measured walkway as quickly as he safely can. Time was recorded to one tenth of a second with a stop watch from when his first foot crossed the start line until when the second foot crossed the finish line. How often the participant , touched the wall was to be noted. Care was taken to ensure that the participants were safe when completing this test. The assessor was allowed to walk nearby to provide 'emergency' help if needed, but must not support or provide manual assistance for the participant in any way. If the participant was unable to complete the 10-meter walk, the total distance was recorded. The participants were to perform the test in bare feet. No aids or orthoses were allowed. Change from Baseline, was defined as the post-randomization value minus the Baseline value. Baseline was defined as Week 0.
Time Frame: Baseline (Week 0) and Week 24
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 16 | 17 | 18
Seconds | -0.04 (0.196) | 0.52 (0.187) | -0.01 (0.185)
Statistical Analysis 1: Comparison: Placebo (Combined) vs GSK2402968 3 mg/kg/Week; Treatment difference: Placebo Vs GSK2402968 3 mg; Test type: Superiority or Other; p = 0.050, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Model included terms for treatment, centre grouping and baseline; Median Difference (Net) = 0.564, 95% CI 2-sided [0.000 to 1.127]
Statistical Analysis 2: Comparison: Placebo (Combined) vs GSK2402968 6 mg/kg/Week; Treatment difference: Placebo Vs GSK2402968 6 mg; Test type: Superiority or Other; p = 0.890, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Model included terms for treatment, center grouping and baseline; Mean Difference (Net) = 0.037, 95% CI 2-sided [-0.498 to 0.571]

5. Secondary Outcome: Change From Baseline in Muscle Strength Total Score at Week 24
Description: The muscle strength was recorded by handheld myometry using a microFET2 myometer. Upper and lower limb proximal muscles were evaluated including knee flexors, knee extensors, elbow flexors, elbow extensors, shoulder abductors and hip flexors. Total score was calculated by summing up all individual scores. If data for any of the individual muscle strength tests was missing, the total score were set to missing for that visit. Change from Baseline, was defined as the post-randomization value minus the Baseline value. Baseline was defined as Week 0.
Time Frame: Baseline (Week 0) and Week 24
Population: ITT Population. Only those participants available at the specified timepoints were analyzed
Measure: Least Squares Mean (Standard Error); unit: Pounds (lbs)
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 16 | 17 | 17
Pounds (lbs) | 0.32 (4.633) | 2.67 (4.385) | 1.14 (4.469)
Statistical Analysis 1: Comparison: Placebo (Combined) vs GSK2402968 3 mg/kg/Week; Treatment difference: Placebo Vs GSK2402968 3 mg; Test type: Superiority or Other; p = 0.723, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Model includes terms for Treatment, Centre Grouping and Baseline Muscle Strength Total Score; Mean Difference (Net) = 2.356, 95% CI 2-sided [-10.936 to 15.648]
Statistical Analysis 2: Comparison: Placebo (Combined) vs GSK2402968 6 mg/kg/Week; Treatment difference: Placebo Vs GSK2402968 6mg; Test type: Superiority or Other; p = 0.898, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Model includes terms for Treatment, Centre Grouping and Baseline Muscle Strength Total Score; Mean Difference (Net) = 0.821, 95% CI 2-sided [-12.034 to 13.676]

6. Secondary Outcome: Change From Baseline in Muscle Strength Tests For-Knee Extensor, Knee Flexor, Hip Flexor, Elbow Flexor, Elbow Extensor, Shoulder Abductor at Week 24
Description: The muscle strength was recorded by handheld myometry using a microFET2 myometer. Upper and lower limb proximal muscles were evaluated including knee flexors, knee extensors, elbow flexors, elbow extensors, shoulder abductors and hip flexors. Change from Baseline, was defined as the post-randomization value minus the Baseline value. Baseline was defined as Week 0.
Time Frame: Baseline (Week 0) and Week 24
Population: ITT population.
Measure: Mean (Standard Deviation); unit: lbs
Groups:
- GSK2402968 3 mg/kg/Week: The participants in this arm were administered with 3 mg per kilogram kg GSK2402968, subcutaneously for 24 weeks. It was provided as 3 mL vials containing 1 mL sterile solution. The concentration of drisapersen solution was 200 mg per mL
- GSK2402968 6 mg/kg/Week: The participants in this arm were administered with 6 mg per kg GSK2402968, subcutaneously for 24 weeks. It was provided as 3 mL vials containing 1 mL sterile solution. The concentration of drisapersen solution was 200 mg per mL
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 16 | 17 | 18
lbs
  Knee extensor left | 0.01 (4.574) | -1.14 (3.219) | 1.02 (3.863)
  Knee extensor right | -0.99 (3.625) | -0.88 (3.123) | 0.45 (3.235)
  Knee flexor left: number analyzed (Participants) | 16 | 17 | 17
  Knee flexor left | 0.10 (3.398) | 0.37 (2.178) | 0.48 (2.211)
  Knee flexor right: number analyzed (Participants) | 16 | 17 | 17
  Knee flexor right | 0.11 (2.763) | 0.05 (2.410) | 0.28 (2.039)
  Hip flexor left: number analyzed (Participants) | 16 | 17 | 17
  Hip flexor left | -0.53 (2.922) | -0.58 (2.848) | 1.10 (3.391)
  Hip flexor right: number analyzed (Participants) | 16 | 17 | 17
  Hip flexor right | -0.82 (4.190) | -0.08 (3.213) | 0.57 (3.243)
  Elbow flexor left | 0.86 (2.443) | 0.56 (2.410) | 0.69 (2.273)
  Elbow flexor right | 0.47 (2.633) | -0.25 (1.737) | 0.11 (1.801)
  Elbow extensor left | 0.50 (1.344) | 0.45 (2.235) | 0.56 (2.547)
  Elbow extensor right | 0.69 (1.673) | 1.11 (2.118) | 0.15 (1.715)
  Shoulder abductor left | 0.13 (1.423) | 0.65 (1.825) | 0.31 (1.710)
  Shoulder abductor right | 0.29 (1.588) | 0.26 (2.150) | 0.69 (2.106)

7. Secondary Outcome: Change From Baseline in the North Star Ambulatory Assessment (NSAA) Total Score
Description: The NSAA was a functional scale devised from Hammersmith Scale of Motor Ability specifically for use in ambulant children with DMD. It consists of 17 activities graded 0 (unable to perform), 1 (performs with modifications), 2 (normal movement). The scale assessed activities that required for ambulatory activity and included items that were rarely achieved in untreated DMD (jump, hop, raise head) as well as items that are known to progressively deteriorate over time (stand from a chair, walk). A standardized manual is available within the SPM with specific instructions for grading. Video snaps used in training program to ensure evaluator reliability. The total score ranged from 0-34 where the highest score of 34 implies absence of symptoms and lower score implies more severe symptoms. Change from Baseline, was defined as the post-randomization value minus the baseline value. Baseline was defined as Week 0.
Time Frame: Baselie (Week 0) and Week 24
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 16 | 17 | 18
Scores on scale | -0.6 (0.84) | -1.1 (0.80) | -0.8 (0.79)
Statistical Analysis 1: Comparison: Placebo (Combined) vs GSK2402968 3 mg/kg/Week; Treatment difference: Placebo Vs GSK2402968 3 mg; Test type: Superiority or Other; p = 0.684, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Model included terms for treatment, center grouping and baseline; Mean Difference (Net) = -0.49, 95% CI 2-sided [-2.90 to 1.92]
Statistical Analysis 2: Comparison: Placebo (Combined) vs GSK2402968 6 mg/kg/Week; Treatment difference: Placebo Vs GSK2402968 6 mg; Test type: Superiority or Other; p = 0.873, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Model included terms for treatment, center grouping and baseline; Mean Difference (Net) = -0.18, 95% CI 2-sided [-2.49 to 2.12]

8. Secondary Outcome: Number of Participants With Accidental Falls During 6 Minute Walk Distance Test
Description: The participants during the 6 minute walk distance were asked to walk, at their own preferred speed, up and down a fixed distance until they were told to stop after 6 minutes. The participants were warned of the time and were told to stop earlier if they feel unable to continue. The total distance walked within the duration of 6 minutes (or until the participant stopped in case of early termination of the test), was recorded in metersThe number of accident falls during the 6 minute walk distance were reported. Data is reported for the number of participants with accidental falls of 0, 1 and 2.
Time Frame: Baseline (Week 0), Week 24, Week 36 and Week 48
Population: ITT Population. Only those participants available at the specified timepoints were analyzed
Measure: Number; unit: Participants
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 16 | 17 | 18
Participants
  Baseline, 0 fall | 16 | 16 | 17
  Baseline, 1 fall | 0 | 1 | 1
  Week 12, 0 fall | 15 | 17 | 17
  Week 12, 1 fall | 1 | 0 | 1
  Week 24, 0 fall | 16 | 16 | 16
  Week 24, 1 fall | 0 | 1 | 2
  Week 36, 0 fall: number analyzed (Participants) | 14 | 14 | 14
  Week 36, 0 fall | 14 | 13 | 14
  Week 36, 2 falls: number analyzed (Participants) | 14 | 14 | 14
  Week 36, 2 falls | 0 | 1 | 0
  Week 48, 0 fall: number analyzed (Participants) | 11 | 14 | 13
  Week 48, 0 fall | 10 | 14 | 13
  Week 48, 3 falls: number analyzed (Participants) | 11 | 14 | 13
  Week 48, 3 falls | 1 | 0 | 0

9. Secondary Outcome: Change From Baseline in Creatinine Kinase Serum Concentrations
Description: Creatine kinase (CK) is a muscle-specific enzyme; its level in plasma is considered to reflect the extent of muscle damage. In the blood samples drawn to this purpose, the plasma level of CK was measured. Change from Baseline, was defined as the post-randomization value minus the baseline value. Baseline was defined as Week 0.
Time Frame: Baseline (Week 0) and Week 48
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: International units per liter
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 16 | 17 | 18
International units per liter
  Week 24: number analyzed (Participants) | 16 | 17 | 17
  Week 24 | -3303.5 (1224.65) | -4196.4 (1171.20) | -4609.0 (1170.75)
  Week 48: number analyzed (Participants) | 15 | 17 | 18
  Week 48 | -2783.1 (1248.65) | -4838.0 (1170.75) | -2615.7 (1149.44)
Statistical Analysis 1: Comparison: Placebo (Combined) vs GSK2402968 3 mg/kg/Week; Treatment difference: Placebo Vs GSK2402968 3 mg, Week 24; Test type: Superiority or Other; p = 0.610, Mixed Model Repeated Measures — [p-value comment as in outcome 2, analysis 1]; Model included terms for treatment, visit, treatment by visit, center grouping, baseline and baseline by visit; Mean Difference (Net) = -892.88, 95% CI 2-sided [-4391.10 to 2605.35]
Statistical Analysis 2: Comparison: Placebo (Combined) vs GSK2402968 3 mg/kg/Week; Treatment difference: Placebo Vs GSK2402968 3 mg, Week 48; Test type: Superiority or Other; p = 0.248, Mixed Model Repeated Measures — [p-value comment as in outcome 2, analysis 1]; Model included terms for treatment, visit, treatment by visit, center grouping, baseline and baseline by visit; Mean Difference (Net) = -2054.86, 95% CI 2-sided [-5587.33 to 1477.60]
Statistical Analysis 3: Comparison: Placebo (Combined) vs GSK2402968 6 mg/kg/Week; Treatment difference: Placebo Vs GSK2402968 6 mg, Week 24; Test type: Superiority or Other; p = 0.439, Mixed Model Repeated Measures — [p-value comment as in outcome 2, analysis 1]; Model included terms for treatment, visit, treatment by visit, center grouping, baseline and baseline by visit; Mean Difference (Net) = -1305.46, 95% CI 2-sided [-4668.41 to 2057.48]
Statistical Analysis 4: Comparison: Placebo (Combined) vs GSK2402968 6 mg/kg/Week; Treatment difference: Placebo Vs GSK2402968 6 mg, Week 48; Test type: Superiority or Other; p = 0.921, Mixed Model Repeated Measures — [p-value comment as in outcome 2, analysis 1]; Model included terms for treatment, visit, treatment by visit, center grouping, baseline and baseline by visit; Mean Difference (Net) = 167.39, 95% CI 2-sided [-3208.98 to 3543.77]

10. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in the First Second of Exhalation (FEV1) at Week 24
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Change from Baseline, was defined as the post-randomization value minus the Baseline value. Baseline was defined as Week 0.
Time Frame: Baseline (Week 0) and Week 24
Population: ITT Population. Only those participants available at the indicated timepoints were used for analysis
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 16 | 16 | 15
Litres | 0.054 (0.2445) | -0.009 (0.2316) | 0.015 (0.1647)

11. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Week 24
Description: FVC is defined as the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Change from Baseline, was defined as the post-randomization value minus the baseline value. Baseline was defined as Week 0.
Time Frame: Baseline (Week 0) and Week 24
Population: ITT population. Only those participants available at the indicated timepoints were used for analysis.
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 16 | 16 | 15
Litres | 0.063 (0.2670) | 0.080 (0.2064) | 0.051 (0.1419)

12. Secondary Outcome: Change From Baseline in Peak Cough Flow at Week 24
Description: The peak cough flow was conducted using a spirometer. Change from Baseline, was defined as the post-randomization value minus the Baseline value. Baseline was defined as Week 0.
Time Frame: Baseline (Week 0) and Week 24
Population: ITT population. Only those participants available at the indicated timepoints were used for analysis
Measure: Mean (Standard Deviation); unit: Litres per minute
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 15 | 15 | 17
Litres per minute | 16.5 (19.03) | 18.2 (24.19) | 18.0 (28.09)

13. Secondary Outcome: Change From Baseline in Peak Expiratory Flow at Week 24
Description: The peak expiratory flow is a measure of the amount of air that can be pushed through the airways in a single rapid exhalation. The peak expiratory flow was measured using spirometry. Change from Baseline, was defined as the post-randomization value minus the baseline value. Baseline was defined as Week 0.
Time Frame: Baseline (Week 0) and Week 24
Population: ITT population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Litres per minute
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 16 | 16 | 17
Litres per minute | 18.9 (35.89) | 2.5 (35.98) | 6.6 (34.68)

14. Secondary Outcome: Change From Baseline in Sniff Pressure Test at Week 24
Description: This was one of the pulmonary function test which was a non-invasive procedure. It measured the inspiratory muscle strength by transdiaphragmatic (Pdi) and esophageal pressures (Pes) generated during volitional and nonvolitional maneuvers. Change from Baseline, was defined as the post-randomization value minus the baseline value. Baseline was defined as Week 0.
Time Frame: Baseline (Week 0) and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Centimeter of water
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 16 | 15 | 16
Centimeter of water | 3.46 (12.988) | -1.47 (10.155) | 2.75 (16.838)

15. Secondary Outcome: Number of Participants With Change From Baseline in Dystrophin Expression at Week 24 by Immunofluorescence Assay (IFA)
Description: A muscle biopsy from the tibialis anterior muscle was taken to assess the expression of dystrophin. The muscle biopsy samples were collected by open biopsy or with the conchotome method according to standard hospital procedures for obtaining muscle biopsies from children. The minimum amount of muscle tissue required is a small piece of muscle of at least 0.5 x 0.5 x 0.5 centimeters. The muscle tissue was immediately frozen in liquid nitrogen-cooled 2-methylbutane and stored at -80°Celsius (C) or -70°C till shipment. In case of DMD participants , there is defect in the dystrophin producing gene or absence. Data for number of participants with change from baseline in dystrophin expression, was diagnosed using IFA and was categorized as strong increase, increase, and no change, decrease.
Time Frame: Baseline (Week 0) and Week 24
Population: ITT population. Only those participants available at the specified timepoints were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 12 | 11 | 13
Participants
  Strong increase | 5 | 3 | 0
  Increase | 2 | 2 | 1
  Decrease | 2 | 3 | 4
  No change | 3 | 3 | 8

16. Secondary Outcome: Number of Clinician Global Impression of Improvement (CGI-I) Responders
Description: Single item question designed to provide a brief, stand-alone assessment of the clinician's view of the participant's global functioning after initiating a study medication, compared to their global functioning just prior to initiating treatment. Evaluated by an expert physician or evaluator familiar with DMD and who could make an expert clinical global judgement about severity of illness across various time points within context of clinical experience. The CGI-I reflects the clinician's judgment about the total picture of the participant : the illness severity, the level of distress and other aspects of impairment, and impact of illness on functioning. The CGI-I is rated without regard to clinician's belief that any clinical changes are or are not due to medication and without consideration of etiology of symptoms. It is measured on 7-point Likert scale (1 = 'very much improved', 2 = 'much improved', 4 = 'no change', 5 = 'minimally worse', 6 = 'much worse', 7 = 'very much worse').
Time Frame: Week 24 and Week 48
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 16 | 17 | 18
Participants
  Week 24: number analyzed (Participants) | 14 | 17 | 18
  Week 24 | 2 | 1 | 2
  Week 48: number analyzed (Participants) | 14 | 17 | 16
  Week 48 | 1 | 0 | 2
Statistical Analysis 1: Comparison: Placebo (Combined) vs GSK2402968 3 mg/kg/Week; Placebo (combined), GSK2402968 3 mg/kg/week; Test type: Superiority or Other; p = 0.541, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Model includes terms for Treatment and Centre Grouping; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.02 to 7.01]
Statistical Analysis 2: Comparison: Placebo (Combined) vs GSK2402968 6 mg/kg/Week; Placebo (combined), GSK2402968 6 mg/kg/week; Test type: Superiority or Other; p = 0.417, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Model includes terms for Treatment and Centre Grouping; Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.03 to 4.27]

17. Secondary Outcome: Assessment of Functional Outcome by : Functional Outcomes Survey During Treatment Period
Description: This was conducted by the family or caregiver. This helped to document the observed changes in the participant's functional outcome like the day to day activities; general health, mobility, and other general daily activities. The data for Week 24 has been reported as improved, not improved and not applicable.
Time Frame: Up to Week 24
Population: ITT population. Only those participants available at that particular time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 16 | 17 | 18
Participants
  Ability to walk 50 feet, improved | 4 | 4 | 8
  Ability to walk 50 feet, not improved | 12 | 13 | 10
  Ability to walk 50 feet, not applicable | 0 | 0 | 0
  Rate your child's condition, improved | 5 | 6 | 6
  Rate your child's condition, not improved | 11 | 11 | 12
  Walk 15-20 mins without tired,improved | 5 | 5 | 6
  Walk 15-20 mins without tired,not improved | 11 | 11 | 12
  Walk 15-20 mins without tired,not applicable | 0 | 1 | 0
  Able to stand 10 mins without tired, improved | 3 | 4 | 4
  Able to stand 10 mins without tired,not improved | 13 | 13 | 14
  Able to stand 10 mins without tired,not applicable | 0 | 0 | 0
  Able to step up on stool, improved | 3 | 5 | 5
  Able to step up on stool, not improved | 13 | 11 | 13
  Able to step up on stool, not applicable | 0 | 1 | 0
  Able to walk up/down a slope, improved | 4 | 5 | 6
  Able to walk up/down a slope, not improved | 11 | 12 | 12
  Able to walk up/down a slope, not applicable | 1 | 0 | 0
  Able to climb 3-4 steps, improved | 2 | 5 | 5
  Able to climb 3-4 steps, not improved | 14 | 12 | 13
  Able to climb 3-4 steps, not applicable | 0 | 0 | 0
  Able to climb 10-15 steps, improved | 2 | 2 | 3
  Able to climb 10-15 steps, not improved | 14 | 14 | 14
  Able to climb 10-15 steps, not applicable | 0 | 1 | 1
  Able to walk on uneven surfaces, improved | 4 | 3 | 5
  Able to walk on uneven surfaces, not improved | 12 | 14 | 13
  Able to walk on uneven surfaces, not applicable | 0 | 0 | 0
  Able to walk without fall, improved | 6 | 5 | 8
  Able to walk without fall, not improved | 10 | 12 | 10
  Able to walk without fall, not applicable | 0 | 0 | 0
  Participate in physical activities, improved | 4 | 3 | 5
  Participate in physical activities, not improved | 12 | 13 | 13
  Participate in physical activities, not applicable | 0 | 1 | 0
  Able to go out with friends/family, improved | 6 | 5 | 5
  Able to go out with friends/family, not improved | 10 | 12 | 12
  Able to go out with friends/family, not applicable | 0 | 0 | 1
  Able to throw and catch ball, improved | 3 | 2 | 6
  Able to throw and catch ball, not improved | 13 | 15 | 12
  Able to throw and catch ball, not applicable | 0 | 0 | 0
  Able to run and kick a ball, improved | 4 | 1 | 6
  Able to run and kick a ball, not improved | 12 | 15 | 12
  Able to run and kick a ball, not applicable | 0 | 1 | 0
  Able to get in and out of bed, improved | 4 | 4 | 6
  Able to get in and out of bed, not improved | 12 | 13 | 11
  Able to get in and out of bed, not applicable | 0 | 0 | 1
  Able to get in and out of car, improved | 4 | 3 | 5
  Able to get in and out of car, not improved | 12 | 14 | 12
  Able to get in and out of car, not applicable | 0 | 0 | 1
  Able to pick small item from table, improved | 1 | 2 | 4
  Able to pick small item from table, not improved | 15 | 15 | 13
  Able to pick small item from table, not applicable | 0 | 0 | 1
  Able to pick large item from table, improved | 2 | 3 | 5
  Able to pick large item from table, not improved | 14 | 14 | 13
  Able to play with toys, improved | 1 | 4 | 3
  Able to play with toys, not improved | 14 | 13 | 13
  Able to play with toys, not applicable | 1 | 0 | 2
  Able to play board or video games, improved | 4 | 4 | 7
  Able to play board or video games, not improved | 12 | 13 | 11
  Able to play board or video games, not applicable | 0 | 0 | 0
  Able to work on computer, improved | 3 | 2 | 4
  Able to work on computer, not improved | 13 | 15 | 12
  Able to work on computer, not applicable | 0 | 0 | 2
  Able to squeeze out toothpaste, improved | 1 | 2 | 3
  Able to squeeze out toothpaste, not improved | 15 | 12 | 14
  Able to squeeze out toothpaste, not applicable | 0 | 3 | 1
  Able to brush teeth, improved | 2 | 2 | 4
  Able to brush teeth, not improved | 14 | 15 | 13
  Able to brush teeth, not applicable | 0 | 0 | 1
  Pour milk or juice from in a cup , improved | 2 | 0 | 5
  Pour milk or juice from in a cup, not improved | 14 | 16 | 11
  Pour milk or juice from in a cup, not applicable | 0 | 1 | 2
  Able to drink from cup without straw, improved | 2 | 2 | 4
  Able to drink from cup without straw, not improved | 14 | 15 | 13
  Drink from cup without straw, not applicable | 0 | 0 | 1
  Able to button shirt or jacket, improved | 2 | 0 | 6
  Able to button shirt or jacket, not improved | 14 | 16 | 10
  Able to button shirt or jacket, not applicable | 0 | 1 | 2
  Able to zip jacket or pants, improved | 1 | 1 | 4
  Able to zip jacket or pants, not improved | 14 | 16 | 13
  Able to zip jacket or pants, not applicable | 1 | 0 | 1
  Childs need for orthotics, improved | 0 | 0 | 0
  Childs need for orthotics, not improved | 9 | 10 | 5
  Childs need for orthotics, not applicable | 7 | 7 | 13
  Childs need for wheelchair, improved | 1 | 0 | 1
  Childs need for wheelchair, not improved | 6 | 10 | 5
  Childs need for wheelchair, not applicable | 9 | 7 | 12

18. Secondary Outcome: Assessment of Functional Outcome by : Physician Assessment of Daily Living
Description: This was conducted by the physician, which helped to assess and document observed changes in the participant by the physician reported by the participant or his family or caregiver. This was reported as any worsening and any improvement up to week 24.
Time Frame: Week 24 and Week 48
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
Number analyzed (Participants) | 16 | 17 | 18
Participants
  Week 12, Any improvement: number analyzed (Participants) | 16 | 16 | 16
  Week 12, Any improvement | 9 | 6 | 12
  Week 12, Any worsening: number analyzed (Participants) | 16 | 16 | 16
  Week 12, Any worsening | 2 | 1 | 0
  Week 24, Any improvement: number analyzed (Participants) | 15 | 17 | 18
  Week 24, Any improvement | 10 | 8 | 13
  Week 24, Any worsening: number analyzed (Participants) | 15 | 17 | 18
  Week 24, Any worsening | 5 | 3 | 3
  Week 48, Any improvement: number analyzed (Participants) | 10 | 14 | 9
  Week 48, Any improvement | 5 | 5 | 7
  Week 48, Any worsening: number analyzed (Participants) | 10 | 14 | 9
  Week 48, Any worsening | 6 | 6 | 3
  Anytime during study, Any improvement | 12 | 11 | 17
  Anytime during study, Any worsening | 11 | 8 | 6

ADVERSE EVENTS:
Time Frame: Up to Week 48
Description: Safety Population was defined as all participants who received at least one dose of study medication.
Groups:
- GSK2402968 3 mg/kg/Week: The participants in this arm were administered with 3 mg per kg GSK2402968, subcutaneously for 24 weeks. It was provided as 3 mL vials containing 1 mL sterile solution. The concentration of drisapersen solution was 200 mg/mL
Arm/Group | Placebo (Combined) | GSK2402968 3 mg/kg/Week | GSK2402968 6 mg/kg/Week
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 13/16 | 16/17 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Combined) (N=16) | GSK2402968 3 mg/kg/Week (N=17) | GSK2402968 6 mg/kg/Week (N=18)
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Combined) (N=16) | GSK2402968 3 mg/kg/Week (N=17) | GSK2402968 6 mg/kg/Week (N=18)
Injection site erythema (General disorders) | 1 (1) | 10 (63) | 9 (97)
Injection site discolouration (General disorders) | 1 (1) | 5 (19) | 5 (37)
Headache (Nervous system disorders) | 4 (24) | 3 (7) | 2 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 4 (5)
Nasopharyngitis (Infections and infestations) | 2 (3) | 4 (5) | 3 (5)
Procedural pain (Injury, poisoning and procedural complications) | 3 (7) | 1 (1) | 4 (6)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 5 (7)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (2) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (5)
Injection site bruising (General disorders) | 1 (1) | 2 (3) | 3 (5)
Proteinuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (7) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (4) | 0 (0) | 2 (2)
Chromaturia (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Injection site pruritus (General disorders) | 1 (1) | 2 (12) | 1 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (5)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (3)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Injection site haematoma (General disorders) | 2 (2) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (6) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Application site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (4) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Autism spectrum disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Blood fibrinogen decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood immunoglobulin G decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
ECG signs of ventricular hypertrophy (Investigations) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (3)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site oedema (General disorders) | 0 (0) | 0 (0) | 1 (3)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle hypertrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Red blood cells urine (Investigations) | 0 (0) | 1 (2) | 0 (0)
Reticulocyte count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Stitch abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue biting (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.